CLINICAL TRIAL: NCT01092819
Title: Functional Outcome and Recovery After STROKE: The FIRST Trial
Brief Title: A Clinical Trial to Assess the Acute Safety and Functional Outcome and Recovery After STROKE: The FIRST Trial
Acronym: FIRST
Status: Completed | Type: Observational
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP 2988.B
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Stroke
Keywords: acute ischemic stroke, large vessel occlusion, natural history, functional outcome
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- acute ischemic stroke: Patients presenting with symptoms of acute ischemic stroke within 8 hours from symptom onset and with an imaging-defined large cerebral vessel occlusion.
  Interventions: Other: Current standard of care for acute ischemic stroke other than IV rtPA or other IA therapies

INTERVENTIONS:
Other: Current standard of care for acute ischemic stroke other than IV rtPA or other IA therapies — The objective of this study is to determine the natural history of acute ischemic stroke from large vessel thromboembolism in the brain. Patients with current standard of care other than IV rtPA or IA therapies will be studied.

SUMMARY:
Current literature has only limited information on the natural history of acute ischemic stroke from large vessel occlusion in a stroke cohort who presents within 8 hours from symptom onset, particularly on 90 day functional outcome as defined by the mRS. Data from this trial will advance our knowledge on this important topic and may serve as a bench mark for future trials

ELIGIBILITY:
Inclusion Criteria:

* From 18 to 85 years of age.
* Evidence of proximal anterior circulation large vessel occlusion (TIMI 0-1)(TICI 0-1) from CT Angiography. Target vessel occlusion may include the anterior circulation.
* Presented with symptoms consistent with acute ischemic stroke within 8 hours of symptom onset. Patients who presented within 3 hours must be ineligible or refractory to IV rtPA therapy.
* At time of enrollment, neurological deficit resulting in an NIH Stroke Scale (NIHSS) score greater than 10
* Known core infarct volume assessed by CTP, CTA or DWI scans

Exclusion Criteria:

* History of stroke in the past 3 months.
* Pre-existing neurological or psychiatric disease that could confound the study results such as a pre-stroke mRS score greater than 1
* Known severe allergy to contrast media
* Uncontrolled hypertension (defined as systolic blood pressure greater than 185 mmHg or diastolic blood pressure less than 110 mmHg)
* CT evidence of the following conditions before enrollment:

  * Significant mass effect with midline shift
  * Evidence of intracranial hemorrhage
* Treated with endovascular therapy for acute stroke
* Life expectancy less than 90 days
* Participation in another clinical investigation that could confound the evaluation of the study

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with symptoms of acute ischemic stroke within 8 hours from symptom onset and with an imaging-defined large cerebral vessel occlusion and a known infarct volume will be enrolled and followed for 90-days.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Functional outcome at 90 days after presentation as defined by a modified Rankin Score of 0-2. | 90 days after presentation

SECONDARY OUTCOMES:
• Good neurological recovery as defined by a NIHSS score of 0-1 at discharge or a 10-point or more improvement in this scale at discharge. | Discharge and 90 days after presentation
All cause mortality | Dishcharge and 90 days after presentation
Incidence of symptomatic and asymptomatic hemorrhage | Dishcharge and 90 days after presentation

CONTACTS AND LOCATIONS:
Overall Officials: Siu Po Sit, PhD, Study Director — Penumbra Inc.
Locations (3):
- Texas Stroke Institute, Plano, Texas, United States
- China (2):
  - Queen Mary Hospital, Hong Kong, Hong Kong
  - The Prince of Wales Hospital, Shatin, Hong Kong